CLINICAL TRIAL: NCT02434809
Title: Investigation of Respiratory Motion-Corrected Cone-Beam CT and Intratreatment Gating Based on Electromagnetic Transponders to Reduce Target Position Uncertainty in Radiation Treatment of Lung Malignancies
Brief Title: Respiratory Motion-Corrected Cone-Beam CT and Intratreatment Gating Based on Electromagnetic Transponders to Reduce Target Position Uncertainty in Radiation Treatment of Lung Malignancies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-225
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Respiratory Motion-Corrected Cone-Beam CT; Radiation; 14-225
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Patients with lung cancer (Experimental): Physician evaluation of patient setup accuracy will be performed using all available images and adjustments will be made as per standard practice. In addition, a respiration motion-corrected CBCT (daily for SBRT, weekly for standard fractionation) will be used to confirm the accuracy of Calypso-based setup. Patients will return for follow up at 3,6, 9, 12, 15, 18, 21 and 24 months (+/- 4 weeks) following completion of radiation therapy. The following assessments will be performed at these visits: history and physical exam, diagnostic CT chest, and toxicity assessment.
  Interventions: Procedure: Bronchoscopic Implantation; Device: Cone-Beam CT-Guided; Radiation: stereotactic body radiation treatments

INTERVENTIONS:
Procedure: Bronchoscopic Implantation — Calypso transponders
Device: Cone-Beam CT-Guided
Radiation: stereotactic body radiation treatments

SUMMARY:
The first purpose of this study is to test a new computer program that reduces the blurring in the cone-beam CT scan and helps the doctor to better locate the tumor. The investigators want to find out what effects, good and/or bad, that this has on the patient and the way we treat the cancer in the lungs.

The second purpose of this study is to test how well this computer program tracks markers in the images, compared to using radio signals to follow the markers.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of malignancy suitable for thoracic radiation therapy
* Patient is planning to undergo radiation therapy for primary or recurrent malignancies of the lung or metastatic malignancies to the lung.
* Age ≥ 18 years old
* Karnofsky Performance Status ≥ 60%
* At least part of the tumor must be visible as observed in a diagnostic or planning CT.
* Able to have bronchoscopic placement of Calypso transponders as confirmed on a recent (within the past 8 weeks) CT scan.

Exclusion Criteria:

* Patients with clinically significant active infections.
* Bronchiectasis in the region of the intended implantation.
* History of hypersensitivity to nickel.
* Other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical study.
* Deemed unable to safely undergo or tolerate flexible bronchoscopy as per institutional guidelines
* Unable to tolerate anesthesia or sedation
* Enrolled in any other clinical studies the investigator believes to be in conflict with this investigation.
* Female patients who are pregnant or nursing

Exclusion criteria for Calypso transponders:

* Implants in the chest region that contain metal or conductive materials (e.g., metal implants, rods, or plates) which Calypso Medical considers will interfere with the Calypso System's electromagnetic localization.
* Active implanted devices, such as pacemakers, defibrillators, and drug infusion pumps since the effects of the Calypso System operation on these devices are unknown.
* Patients whose lung tumors are being monitored by MR imaging as part of standard clinical care. Implantation of transponders will degrade MR images.
* Posterior lesions that would be >19 cm distance from Calypso detector plate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-04; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
successful Calypso transponder implantation | 1 year
  The RapidTrack algorithm will be considered successful if the centroid position of the Calypso transponders, as determined by the RapidTrack algorithm, are within 2 mm of the positions determined by the Calypso system 95% of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Peng, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/